CLINICAL TRIAL: NCT01278901
Title: The Effect of PPI Therapy on the Result of Helicobacter Pylori Diagnostic Tests
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Vered Shabat, MD, RMC
Other Study IDs: 20100300
Record Dates: First submitted 2011-01-16; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Helicobacter Pylori
Keywords: helicobacter pylori; urease test; 13C-UBT; the focus of the study is to evaluate a possible effect of PPI therapy on Helicobacter pylori diagnostic tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort of consecutive patients undergoing EGD treated with PPI: Patients positive for helicobacter pylori undergoing EGD, started on PPI therapy for a month, repeated diagnostic tests for Helicobacter pylori after a month of therapy (urease test, histology and breath test)

SUMMARY:
STUDY PROTOCOL:

The study will include 30 patients ages 18-80y that had a gastroscopy for various reasons. The patients should not be on PPI therapy . If during the gastroscopy there are some pathologies that require a second look endoscopy after some weeks of therapy (ulcers or esophagitis), the investigators will repeat the gastroscopy within a month.

During the first gastroscopy a biopsy will be taken for histological examination and for a rapid urease test and an urea breath test will be done soon after the procedure.

If one of the tests is positive the investigators postulate that the Helicobacter pylori is actually present.

After the gastroscopy the patient is given a full dose of PPI (as indicated) and helicobacter tests are repeated in the next endoscopy (under PPI therapy) . Any positive test that become negative in the second endoscopy is considered false negative.

ELIGIBILITY:
Inclusion Criteria:

* Cohort of helicobacter pylori positive patients undergoing EGD for different indications and not treated with PPI-

Exclusion Criteria:

* Patients younger than 18 years and older than 80 years
* Severe background diseases
* Previous eradicated helicobacter pylori infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of helicobacter pylori positive patients undergoing EGD for different indications and not treated with PPI
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Effect of PPI treatment on helicobacter pylori diagnostic tests | 1 month of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Rabin Medical Center, Petah Tikva, Israel